CLINICAL TRIAL: NCT00861757
Title: A Phase 3, Randomized, Double Blind, Placebo and Tamsulosin Controlled, Parallel Design, Multinational Study to Evaluate the Efficacy and Safety of Tadalafil Once a Day Dosing for 12 Weeks in Asian Men With Signs and Symptoms of Benign Prostatic Hyperplasia
Brief Title: Multinational Study to Evaluate Tadalafil in Asian Men With Signs and Symptoms of Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10487; H6D-MC-LVHB (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Results first posted 2011-06-13 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tadalafil; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- 2.5 mg Tadalafil (Experimental)
  Interventions: Drug: Tadalafil
- 5.0 mg Tadalafil (Experimental)
  Interventions: Drug: Tadalafil
- 0.2 mg Tamsulosin (Active Comparator)
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tadalafil — by mouth (PO), once daily (QD) (30 min after meal) for 12 weeks
  Other Names: LY450190, Cialis
  Arms: 2.5 mg Tadalafil; 5.0 mg Tadalafil
Drug: Placebo — PO, QD (30 min after meal) for 12 weeks
  Arms: Placebo
Drug: Tamsulosin — PO, QD (30 min after meal) for 12 weeks
  Arms: 0.2 mg Tamsulosin

SUMMARY:
This study is a randomized, double-blind, placebo and tamsulosin-controlled, parallel design, multinational study to evaluate the efficacy and safety of Tadalafil once-a-day dosing for 12 weeks in Asian men with signs and symptoms of benign prostatic hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

* Asian males, with benign prostatic hyperplasia (BPH) for at least 6 months prior to initiation and IPSS score greater than or equal to 13 at the beginning of the treatment
* Agree not to use any other approved or experimental pharmacologic BPH, erectile dysfunction (ED) and overactive bladder (OAB) treatments at any time during the study.
* Have not taken Finasteride or Dutasteride therapy, Anti-androgenic hormone or any other BPH therapy, ED or OAB therapy for specified duration of time prior to the beginning of the treatment

Exclusion Criteria:

* Prostate specific antigen (PSA) score beyond acceptable range defined for study at initiation
* History of urinary retention or lower urinary tract (bladder) stones within 6 months of initiation
* History of urinary urethral obstruction due to stricture, valves, sclerosis, or tumor at initiation
* Clinical evidence of prostate cancer at initiation
* Clinical evidence of any of the bladder or urinary tract conditions, which may affect lower urinary tract symptom at initiation
* History of cardiac conditions, including Angina requiring certain treatment with nitrates, unstable angina defined for study, positive cardiac stress test before starting the study
* History of significant central nervous system injuries (including stroke or spinal cord injury within 6 months of initiation)
* Use of any nitrates, cancer chemotherapy, androgens, antiandrogens, estrogens, luteinizing hormone-releasing hormone (LHRH)agonists/antagonists, or anabolic steroids at initiation

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- Japan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- Taiwan (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kaohsiung City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taoyuan District

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Drug: Placebo by mouth (PO), once daily (QD) (30 min after meal) for 12 weeks
- 2.5 mg Tadalafil; 5.0 mg Tadalafil: Drug: Tadalafil PO, QD (30 min after meal) for 12 weeks
- 0.2 mg Tamsulosin: Drug: Tamsulosin PO, QD (30 min after meal) for 12 weeks
Period: Overall Study
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 0.2 mg Tamsulosin
Started | 154 | 151 | 155 | 152
Completed | 145 | 136 | 137 | 143
Not Completed | 9 | 15 | 18 | 9
Not completed — Adverse Event | 1 | 5 | 7 | 2
Not completed — Entry Criteria Not Met | 1 | 2 | 1 | 1
Not completed — Lack of Efficacy | 3 | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 2 | 4 | 1
Not completed — Withdrawal by Subject | 1 | 5 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 0.2 mg Tamsulosin | Total
Number analyzed (Participants) | 154 | 151 | 155 | 152 | 612
Age Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.1) | 63.7 (7.2) | 62.3 (8.0) | 62.6 (7.9) | 63.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 154 | 151 | 155 | 152 | 612
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 154 | 151 | 155 | 152 | 612
Region of Enrollment [Number; unit: participants]
  Taiwan | 24 | 23 | 21 | 22 | 90
  Japan | 86 | 84 | 87 | 85 | 342
  Korea, Republic of | 44 | 44 | 47 | 45 | 180
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/square meters (kg/m^2)] — Body mass index is an estimate of body fat based on body weight divided by height squared.
  kilograms/square meters (kg/m^2) | 24.3 (2.9) | 23.9 (2.8) | 24.2 (2.8) | 24.4 (2.9) | 24.2 (2.8)
Current Tobacco Use [Number; unit: participants]
  Yes | 27 | 30 | 36 | 23 | 116
  No | 127 | 121 | 119 | 129 | 496
Current Alcohol Use [Number; unit: participants]
  Yes | 78 | 81 | 84 | 83 | 326
  No | 76 | 70 | 71 | 69 | 286
Benign Prostatic Hyperplasia (BPH) Severity [Number; unit: participants] — The International Prostate Symptom Score (IPSS) Total Score is obtained by combining the scores of the responses to 1 through 7 component questions. Each question is scored from 0-5 for an IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
  participants
    Moderate (IPSS<20) | 102 | 102 | 102 | 102 | 408
    Severe (IPSS>=20) | 52 | 49 | 53 | 50 | 204
Duration of BPH [Mean (Standard Deviation); unit: Years] | 3.7 (3.4) | 3.7 (3.3) | 3.5 (2.9) | 3.7 (3.2) | 3.7 (3.2)
Patient Global Impressions of Severity Scale (PGI-S) [Number; unit: participants] — The Patient Global Impressions of Severity Scale (PGI-S) measures patient's perception of severity of illness prior to clinical assessments during study visits. Scores range from 1 (Normal) to 4 (Severe) where 1=Normal, 2=Mild, 3=Moderate, and 4=Severe.
  participants
    Normal | 2 | 0 | 0 | 0 | 2
    Mild | 45 | 41 | 43 | 39 | 168
    Moderate | 92 | 92 | 100 | 93 | 377
    Severe | 15 | 18 | 12 | 20 | 65
Clinical Global Impressions of Severity Scale (CGI-S) [Number; unit: participants] — The Clinical Global Impressions of Severity Scale (CGI-S) measures clinician's perception of severity of illness prior to assessments during study visits. Scores range from 1 (Normal) to 4 (Severe) where 1=Normal, 2=Mild, 3=Moderate, and 4=Severe.
  participants
    Normal | 1 | 0 | 0 | 0 | 1
    Mild | 42 | 36 | 33 | 35 | 146
    Moderate | 97 | 87 | 95 | 92 | 371
    Severe | 14 | 28 | 27 | 25 | 94
Previous Alpha-Blocker Therapy [Number; unit: participants]
  Yes | 83 | 83 | 82 | 87 | 335
  No | 71 | 68 | 73 | 65 | 277
Previous BPH Therapy [Number; unit: participants]
  Yes | 28 | 28 | 36 | 27 | 119
  No | 126 | 123 | 119 | 125 | 493
Postvoid Residual Volume (PVR) [Mean (Standard Deviation); unit: milliliters (mL)] — Postvoid residual volume (PVR) is defined as the volume of urine remaining in the bladder after voiding, estimated by ultrasound.
  milliliters (mL) | 41.9 (47.7) | 37.7 (40.3) | 38.4 (51.2) | 32.7 (37.1) | 37.7 (44.5)
Prostate Volume [Mean (Standard Deviation); unit: mL] — Prostate volume is defined as the volume of prostate estimated by transabdominal or transrectal ultrasound.
  mL | 35.1 (14.0) | 35.3 (16.1) | 34.8 (13.7) | 33.9 (11.1) | 34.8 (13.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) at 12 Weeks
Description: The IPSS Total Score is obtained by combining the scores of the responses to 1 through 7 component questions. Each question is scored from 0-5 for an IPSS range of 0-35 points; higher numerical scores from the IPSS questionnaire represent greater severity of symptoms.
  Least Squares Mean values were controlled for prior alpha blocker use (yes/no), country (Japan/Korea/Taiwan) and baseline value.
Time Frame: baseline, 12 weeks
Population: The primary analysis population for efficacy included all subjects who were randomized and started study medication. All efficacy analyses were performed on an intent-to-treat (ITT) basis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Placebo: Drug: Placebo PO, QD (30min after meal) for 12 weeks
- 2.5 mg Tadalafil; 5 mg Tadalafil: Drug: Tadalafil PO, QD (30min after meal) for 12 weeks
- 0.2 mg Tamsulosin: Drug: Tamsulosin PO, QD (30min after meal) for 12 weeks
Arm/Group | Placebo | 2.5 mg Tadalafil | 5 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 154 | 151 | 154 | 152
Units on a scale | -3.0 (0.4) | -4.8 (0.4) | -4.7 (0.4) | -5.5 (0.4)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-3.0 to -0.6], Standard Error of Mean 0.6
Statistical Analysis 2: Comparison: Placebo vs 5 mg Tadalafil; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = -1.7, 95% CI 2-sided [-2.9 to -0.6], Standard Error of Mean 0.6
Statistical Analysis 3: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -2.5, 95% CI 2-sided [-3.7 to -1.3], Standard Error of Mean 0.6

2. Secondary Outcome: Change From Baseline to 12 Weeks in International Prostate Symptom Score (IPSS) Subscore (Storage [Irritative] and Voiding [Obstructive])
Description: IPSS obstructive subscore is the sum of Questions 1, 3, 5 and 6 of the IPSS questionnaire. Scores range from 0 (few obstructive symptoms) to 5 (frequent obstructive symptoms); 4 questions of the obstructive score range from 0 to 20. IPSS irritative subscore is the sum of Questions 2, 4 and 7 of IPSS questionnaire. Scores range from 0 (no irritative symptoms) to 5 (frequent irritative symptoms); 3 questions of the irritative subscore range from 0 to 15. Least Squares Mean values were controlled for prior alpha blocker use (yes/no), country (Japan/Korea/Taiwan), and baseline value.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 154 | 151 | 154 | 152
units on a scale
  Voiding (Obstructive) Score (N = 154,151,155,152) | -1.9 (0.3) | -3.3 (0.3) | -3.0 (0.3) | -3.8 (0.3)
  Storage (Irritative) Score (N = 154,151,155,152) | -1.1 (0.2) | -1.5 (0.2) | -1.7 (0.2) | -1.7 (0.2)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p < 0.001, ANCOVA — This is the p value for the Voiding (Obstructive) Score; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-2.2 to -0.6], Standard Error of Mean 0.4
Statistical Analysis 2: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p = 0.005, ANCOVA — This is the p value for the Voiding (Obstructive) Score; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-1.9 to -0.3], Standard Error of Mean 0.4
Statistical Analysis 3: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p < 0.001, ANCOVA — This is the p value for the Voiding (Obstructive) Score; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-2.7 to -1.1], Standard Error of Mean 0.4
Statistical Analysis 4: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.072, ANCOVA — This is the p value for the Storage (Irritative) Score; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.0 to 0.0], Standard Error of Mean 0.3
Statistical Analysis 5: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p = 0.021, ANCOVA — This is the p value for the Storage (Irritative) Score; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.1 to -0.1], Standard Error of Mean 0.3
Statistical Analysis 6: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p = 0.023, ANCOVA — This is the p value for the Storage (Irritative) Score; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.1 to -0.1], Standard Error of Mean 0.3

3. Secondary Outcome: Change From Baseline in International Prostate Symptom Score (IPSS) Quality of Life (QoL) at 12 Weeks
Description: Assessment of QoL by urinary symptoms, with scores ranging from 0 (delighted) to 6 (terrible).
  Least Squares Mean values were controlled for Benign Prostatic Hyperplasia severity (moderate/severe), prior alpha blocker use (yes/no), country (Japan/Korea/Taiwan), and baseline value.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 154 | 151 | 154 | 152
units on a scale | -0.5 (0.1) | -0.8 (0.1) | -0.8 (0.1) | -1.1 (0.1)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.031, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to -0.0], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p = 0.013, ANCOVA; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.6 to -0.1], Standard Error of Mean 0.1
Statistical Analysis 3: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.9 to -0.4], Standard Error of Mean 0.1

4. Secondary Outcome: Change From Baseline in Benign Prostatic Hyperplasia (PBH) Impact Index (BII) at 12 Weeks
Description: The BII is a 4-item, self-administered questionnaire evaluating impact of urinary problems on overall health and activity. Total scores range from 0 to 13; higher scores represent increased perceived impact of benign prostatic hyperplasia-lower urinary tract symptoms on overall health. Least Squares Mean values were controlled for BPH severity (moderate/severe), prior alpha blocker use (yes/no), country (Japan/Korea/Taiwan) and baseline value.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 152 | 147 | 153 | 150
units on a scale | -0.8 (0.2) | -1.1 (0.2) | -1.0 (0.2) | -1.6 (0.2)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.201, ANCOVA; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.0 to 0.2], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p = 0.393, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.8 to 0.3], Standard Error of Mean 0.3
Statistical Analysis 3: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p = 0.007, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.4 to -0.2], Standard Error of Mean 0.3

5. Secondary Outcome: Change From Baseline in Uroflowmetry Parameter: Peak Flow Rate (Qmax) at 12 Weeks
Description: Qmax: defined as the peak urine flow rate (measured in milliliters per second [mL/second] using standard calibrated flowmeter).
  Least Squares Mean values were controlled for Benign Prostatic Hyperplasia (BPH) severity (moderate/severe), prior alpha blocker use (yes/no), country (Japan/Korea/Taiwan), and baseline value.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milliliter per second (mL/sec)
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 147 | 145 | 148 | 148
milliliter per second (mL/sec) | 2.1 (0.4) | 1.6 (0.4) | 1.3 (0.4) | 2.1 (0.4)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.331, ANCOVA; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.6 to 0.5], Standard Error of Mean 0.5
Statistical Analysis 2: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p = 0.140, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.8 to 0.3], Standard Error of Mean 0.5
Statistical Analysis 3: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p = 0.940, ANCOVA; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-1.1 to 1.0], Standard Error of Mean 0.5

6. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) at Week 12
Description: The PGI-I measures the patient's perception of improvement at the time of assessment compared with the start of treatment. There are 7 categories with scores ranging from 1 (very much better) to 7 (very much worse). The data are presented as the number of participants in each of the 7 categories: very much better (1); much better (2); a little better (3); no change (4); a little worse (5); much worse (6); very much worse (7).
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 154 | 151 | 155 | 152
Participants
  Very Much Worse | 2 | 1 | 1 | 0
  Much Worse | 3 | 1 | 0 | 1
  A Little Worse | 12 | 4 | 5 | 4
  No Change | 45 | 26 | 23 | 25
  A Little Better | 54 | 62 | 74 | 58
  Much Better | 32 | 44 | 40 | 53
  Very Much Better | 4 | 9 | 10 | 9
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The p-value came from the Cochran-Mantel-Haenszel test to assess if there was any association between treatment (that is, placebo vs 2.5 mg Tadalafil) and 7 categories of the PGI-I
Statistical Analysis 2: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The p-value came from the Cochran-Mantel-Haenszel test to assess if there was any association between treatment (that is, placebo vs 5.0 mg Tadalafil) and 7 categories of the PGI-I
Statistical Analysis 3: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — The p-value came from the Cochran-Mantel-Haenszel test to assess if there was any association between treatment (placebo vs 0.2 mg Tamsulosin) and 7 categories of the PGI-I

7. Secondary Outcome: Clinician Global Impression of Improvement (CGI-I) at Week 12
Description: The CGI-I measures clinician's perception of patient improvement at the time of assessment compared with the start of treatment. There are 7 categories with scores ranging from 1 (very much better) to 7 (very much worse). The data are presented as the number of participants in each of the 7 categories: very much better (1); much better (2); a little better (3); no change (4); a little worse (5); much worse (6); very much worse (7).
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 154 | 151 | 155 | 152
participants
  Very Much Worse | 0 | 2 | 0 | 0
  Much Worse | 3 | 3 | 1 | 1
  A Little Worse | 8 | 4 | 3 | 3
  No Change | 44 | 21 | 29 | 19
  A Little Better | 60 | 67 | 62 | 68
  Much Better | 30 | 39 | 48 | 47
  Very Much Better | 7 | 11 | 10 | 12
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.034, Cochran-Mantel-Haenszel — The p-value came from the Cochran-Mantel-Haenszel test to assess if there was any association between treatment (that is, placebo vs 2.5 mg Tadalafil) and 7 categories of the CGI-I
Statistical Analysis 2: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — The p-value came from the Cochran-Mantel-Haenszel test to assess if there was any association between treatment (that is, placebo vs 5.0 mg Tadalafil) and 7 categories of the CGI-I
Statistical Analysis 3: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — The p-value came from the Cochran-Mantel-Haenszel test to assess if there was any association between treatment (that is, placebo vs 0.2 mg Tamsulosin) and 7 categories of the CGI-I

8. Secondary Outcome: Change From Baseline in Prostate Specific Antigen (PSA) at 12 Weeks
Description: Nanograms of PSA per milliliter (ng/mL) of blood.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microgram/Liter
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 152 | 148 | 153 | 150
microgram/Liter | -0.03 (0.55) | 0.04 (0.54) | 0.13 (0.59) | -0.06 (0.61)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.412, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p = 0.083, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p = 0.456, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Change From Baseline in Postvoid Residual Volume (PVR) at 12 Weeks
Description: The PVR is defined as the volume of urine remaining in the bladder after voiding, estimated by ultrasound.
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 152 | 151 | 153 | 152
milliliter (mL) | -1.20 (45.35) | -0.09 (45.21) | -2.90 (48.84) | -5.67 (34.38)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.688, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p = 0.510, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p = 0.212, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Change From Baseline in Blood Pressure (Sitting) at 12 Weeks
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 154 | 151 | 154 | 152
mm Hg
  Systolic Blood Pressure | 0.9 (10.9) | -2.3 (11.0) | -0.5 (12.4) | 0.2 (12.2)
  Diastolic Blood Pressure | -0.3 (8.6) | -2.5 (7.8) | -1.4 (8.1) | -0.6 (7.9)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.005, Wilcoxon (Mann-Whitney) — This is the p value for systolic blood pressure
Statistical Analysis 2: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p = 0.274, Wilcoxon (Mann-Whitney) — This is the p value for systolic blood pressure
Statistical Analysis 3: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p = 0.538, Wilcoxon (Mann-Whitney) — This is the p value for systolic blood pressure
Statistical Analysis 4: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney) — This is the p value for diastolic blood pressure
Statistical Analysis 5: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p = 0.216, Wilcoxon (Mann-Whitney) — This is the p value for diastolic blood pressure
Statistical Analysis 6: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p = 0.524, Wilcoxon (Mann-Whitney) — This is the p value for diastolic blood pressure

11. Secondary Outcome: Change From Baseline in Blood Pressure (Standing) at 12 Weeks
Time Frame: baseline, 12 weeks
Population: All efficacy analyses were performed on an intent-to-treat (ITT) basis. The primary analysis population for efficacy was the Full Analysis Set (FAS) which included all subjects who were randomized and started study medication.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 154 | 151 | 154 | 152
mm Hg
  Systolic Blood Pressure | 0.8 (11.8) | -2.9 (12.3) | 0.6 (11.6) | -0.9 (13.7)
  Diastolic Blood Pressure | 0.4 (8.1) | -2.3 (8.0) | -1.7 (8.2) | -1.0 (8.8)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.007, Wilcoxon rank-sum test — This is the p value for systolic blood pressure
Statistical Analysis 2: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p = 0.723, Wilcoxon rank-sum test — This is the p value for systolic blood pressure
Statistical Analysis 3: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p = 0.273, Wilcoxon rank-sum test — This is the p value for systolic blood pressure
Statistical Analysis 4: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.005, Wilcoxon rank-sum test — This is the p value for diastolic blood pressure
Statistical Analysis 5: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p = 0.054, Wilcoxon rank-sum test — This is the p value for diastolic blood pressure
Statistical Analysis 6: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p = 0.278, Wilcoxon rank-sum test — This is the p value for diastolic blood pressure

12. Secondary Outcome: Change From Baseline in Sitting Heart Rate (HR) at 12 Weeks
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 0.2 mg Tamsulosin
Number analyzed (Participants) | 154 | 151 | 154 | 152
beats per minute (bpm) | -0.3 (8.9) | 0.7 (8.3) | 0.6 (8.3) | 0.6 (7.8)
Statistical Analysis 1: Comparison: Placebo vs 2.5 mg Tadalafil; Test type: Superiority or Other; p = 0.330, Wilcoxon rank-sum test
Statistical Analysis 2: Comparison: Placebo vs 5.0 mg Tadalafil; Test type: Superiority or Other; p = 0.838, Wilcoxon rank-sum test
Statistical Analysis 3: Comparison: Placebo vs 0.2 mg Tamsulosin; Test type: Superiority or Other; p = 0.409, Wilcoxon rank-sum test

ADVERSE EVENTS:
Arm/Group | Placebo | 2.5 mg Tadalafil | 5.0 mg Tadalafil | 0.2 mg Tamsulosin
Serious Adverse Events (participants affected / at risk) | 1/154 | 4/151 | 0/155 | 0/152
Other Adverse Events (participants affected / at risk) | 24/154 | 38/151 | 42/155 | 35/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=154) | 2.5 mg Tadalafil (N=151) | 5.0 mg Tadalafil (N=155) | 0.2 mg Tamsulosin (N=152)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=154) | 2.5 mg Tadalafil (N=151) | 5.0 mg Tadalafil (N=155) | 0.2 mg Tamsulosin (N=152)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reflux oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis A (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Glucose urine present (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Transaminases abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 6 (7) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 3 (4) | 3 (3) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spontaneous penile erection (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon polypectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days